CLINICAL TRIAL: NCT01867359
Title: The Genetic Characterization of Dementia
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903326; 03-AG-N326
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-09-20

CONDITIONS: Dementia
Keywords: Alzheimer Disease; Molecular; Molecular Genetics; DNA
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Background:

- Researchers are interested in learning more about dementia and its causes. They want to look at the genetic basis of dementia. Identifying genetic aspects of dementia may help provide better tests and treatments for it. It may also show rare gene variants that can cause or alter a person's risks for developing dementia. This study will look at people who have dementia, their family members, and healthy volunteers.

Objectives:

- To study genetic influences on dementia.

Eligibility:

* Individuals who have been diagnosed with dementia.
* Family members of individuals who have been diagnosed with dementia.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will be interviewed and answer questions about their medical history. They will also provide general information on the relatives' medical histories.
* Participants will provide a blood sample for genetic testing.
* Participants will remain on the study for up to 10 years. They will have regular visits to monitor their brain health and function.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Dementia is a condition of declining mental abilities, especially memory. Dementia can occur at any age but becomes more frequent with age, with a prevalence of 5%-10% in people over 65 and 20% in people over 80. Dementia affects the rate of information processing, short term memory is affected before long term memory. It is difficult to diagnose between even the three most common types: Alzheimers disease, Lewy Body disease and multi infarct dementia.

Alzheimer's disease (AD) is a genetically complex and heterogeneous disorder. It is the most common form of dementia, accounting for about 50-70% of typical, late onset cases of dementia. To date, mutations in three genes (APP, PSEN1, PSEN2) have been described to cause familial early-onset AD. In addition, a common polymorphism in the gene encoding apolipoprotein E (APOE) has been associated with the more common late-onset form of the disease. Genetic variability at the APOE locus is a major determinant of late onset Alzheimer s disease. Recent estimates suggest that these four established genes account for less than 30% of the genetic variance in age of onset for AD and predict that numerous AD genes may exist.

Lewy Body Disease includes a range of disorders: Parkinson s Disease, Dementia with Lewy bodies, and Parkinson s dementia, among others. Dementia with Lewy bodies (DLB) accounts for 20% of all cases of dementia in old age. Clinically DLB is characterized by cognitive impairment, visual hallucinations, and parkinsonism. Lewy bodies are neuronal inclusions comprised of abnormally truncated and phosphorylated neurofilament proteins, alpha-synuclein, ubiquitin and associated enzymes. Mutations in the alpha synuclein gene were first discovered in 1996 in a family with autosomal dominant Lewy body parkinsonism. However, most lewy body parkinsonism is not due to a variant in the alpha-synuclein gene. The importance of alpha-synuclein is attributed to the finding of antibodies to alpha -synuclein stain Lewy bodies in brains of all Lewy body disease cases. The ability to identify underlying genetic influences that result in different synuclein pathologies is key to understanding these disorders.

The first aim of this protocol is to collect families with a history of dementia in an attempt to clone the causative gene defect(s) via linkage and positional cloning. Our experience with the cloning of the Amyloid Precursor Protein mutations in Alzheimer s disease shows that this approach leads to a better understanding of the biochemical and physiological processes underlying the disease.

It is clear there are numerous forms of dementia where disease does not appear to be inherited in a Mendelian manner. Whilst these may be caused by environmental effects it is also reasonable to hypothesize that disease may be caused by complex genetic interactions. Furthermore, the susceptibility to environmental influence may be affected by genetic predisposition. As a second aim in this protocol, we will investigate the association between genetic polymorphisms and dementia. This will be performed by a candidate gene approach, assessing the contribution of genes already associated with familial forms of disease, likely candidates (for example involved in the cholinergic system, cell survival or Beta Amyloid processing) or genes within a genetic region previously linked to disease. Although significant association does not imply a causal relationship between the presence of the variant and disease, the pathophysiologic significance should be studied further. The inevitable problem of false positives within this type of analysis is a real one, which may be addressed by independent replications and tightly controlled experiments. Undeniably the analytical effort needed to differentiate positives from false positives is considerable, and as can be readily seen in Alzheimer s disease, the literature is scattered with positive associations and subsequent refutations. However, it is important that research groups continue to identify and replicate these studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Previous diagnosis of Dementia by neurologist, other medical care provider, or researcher accompanied by sufficient clinical and/or laboratory evidence

Clinical confirmation of Dementia by the investigator and his associates either by exam and/or review of medical records

Family member of diagnosed dementia patient

Healthy controls

EXCLUSION CRITERIA:

Individuals with any movement disorder secondary to a specific environmental exposure, birth injury, metabolic disorder, or brain infection such as encephalitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2003-03-14; Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20

PRIMARY OUTCOMES:
Genetic cause of disease identified | Once every 12-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Singleton, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States